CLINICAL TRIAL: NCT03720041
Title: Myeloma XIV: A Phase III Trial to Compare Standard and Frailty-adjusted Induction Therapy With Ixazomib, Lenalidomide and Dexamethasone (IRD) and Maintenance Lenalidomide (R) to Lenalidomide Plus Ixazomib (R+I)
Brief Title: Myeloma XIV: Frailty-adjusted Therapy in Transplant Non-Eligible Patients With Newly Diagnosed Multiple Myeloma
Acronym: FiTNEss
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: Cancer Research UK (Other); Takeda (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MyelomaXIV
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2020-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Lenalidomide; Ixazomib; Dexamethasone; Revlimid; Ninlaro; Non-transplant eligible myeloma patients; Newly diagnosed myeloma; Double blind; Placebo; Frailty scoring; Frailty score-adjusted dosing
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; ixazomib

STUDY DESIGN:
Intervention Model Description: Phase III, multi-centre, randomised, parallel group trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation 1 is open label Randomisation 2 is double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- R1: IRD induction therapy (reactive) (Active Comparator): In the reactive arm at Randomisation 1, participants will receive IRD induction therapy with standard up-front dosing, with toxicity assessed at each cycle and doses adjusted in accordance with the guidelines given in the trial protocol.
  Interventions: Drug: R1: Ixazomib, Lenalidomide, Dexamethasone (IRD) induction therapy - reactive arm
- R1: IRD induction therapy (adaptive) (Experimental): In the adaptive arm at Randomisation 1, participants will receive IRD induction therapy with up-front dose reductions adjusted according to their frailty score: fit, unfit, or frail.
  Interventions: Drug: R1: Ixazomib, Lenalidomide, Dexamethasone (IRD) induction therapy - adaptive arm
- R2: Lenalidomide plus placebo maintenance (Active Comparator): Participants randomised to this arm at Randomisation 2 will receive lenalidomide plus placebo maintenance.
  Interventions: Drug: R2: Lenalidomide plus placebo maintenance
- R2: Lenalidomide + ixazomib maintenance (Experimental): Participants randomised to this arm at Randomisation 2 will receive lenalidomide plus ixazomib maintenance.
  Interventions: Drug: R2: Lenalidomide + ixazomib maintenance

INTERVENTIONS:
Drug: R1: Ixazomib, Lenalidomide, Dexamethasone (IRD) induction therapy - reactive arm — In the reactive arm at Randomisation 1, participants will receive IRD induction therapy with standard up-front dosing, with toxicity assessed at each cycle and doses adjusted in accordance with the guidelines given in the trial protocol. All participants will be given the following starting doses:
  Ixazomib: 4mg/day on days 1, 8 and 15, taken orally
  Lenalidomide: 25mg/day on days 1-21, taken orally
  Dexamethasone: 40mg on days 1, 8, 15 and 22 for participants aged ≤75 years, or 20mg on days 1, 8, 15 and 22 for participants aged > 75 years; taken orally
  Participants will receive this dosing regimen for 12 cycles of induction treatment, in the absence of disease progression or unacceptable toxicity. Each cycle is 28 days.
  Other Names: Ninlaro; Revlimid
  Arms: R1: IRD induction therapy (reactive)
Drug: R1: Ixazomib, Lenalidomide, Dexamethasone (IRD) induction therapy - adaptive arm — In the adaptive arm at Randomisation 1, participants will receive IRD induction therapy with up-front dose reductions adjusted according to their frailty score: fit, unfit, or frail. The starting doses for each frailty category are described below:
  1. Fit category:
     Ixazomib: 4mg/day on days 1, 8 and 15, taken orally Lenalidomide: 25mg on days 1-21, taken orally Dexamethasone: 40mg on days 1, 8, 15 and 22, taken orally
  2. Unfit category:
     Ixazomib: 4mg/day on days 1, 8 and 15, taken orally Lenalidomide: 15mg on days 1-21, taken orally Dexamethasone: 20mg on days 1, 8, 15 and 22, taken orally
  3. Frail category:
  Ixazomib: 4mg/day on days 1, 8 and 15, taken orally Lenalidomide: 10mg on days 1-21, taken orally Dexamethasone: 10mg on days 1, 8, 15 and 22, taken orally
  Participants will receive this dosing regimen for 12 cycles of induction treatment, in the absence of disease progression or unacceptable toxicity. Each cycle is 28 days.
  Other Names: Ninlaro; Revlimid
  Arms: R1: IRD induction therapy (adaptive)
Drug: R2: Lenalidomide plus placebo maintenance — Participants randomised to receive lenalidomide plus placebo maintenance at Randomisation 2 will receive the following starting doses:
  Lenalidomide: 10mg*/day on days 1-21, taken orally Placebo: 4mg*/day on days 1, 8 and 15
  * or final dose administered at the end of induction treatment if lower.
  This dosing regimen is continued for every maintenance cycle. Participants will continue maintenance treatment until disease progression or intolerance/unacceptable toxicity. Each maintenance cycle is 28 days.
  Randomisation 2 is double-blind - participants and their treating clinicians will be blinded to maintenance allocation.
  Other Names: Revlimid
  Arms: R2: Lenalidomide plus placebo maintenance
Drug: R2: Lenalidomide + ixazomib maintenance — Participants randomised to receive lenalidomide plus ixazomib maintenance at Randomisation 2 will receive the following starting doses:
  Lenalidomide: 10mg*/day on days 1-21, taken orally Ixazomib: 4mg*/day on days 1, 8 and 15
  * or final dose administered at the end of induction treatment if lower.
  This dosing regimen is continued for every maintenance cycle. Participants will continue maintenance treatment until disease progression or intolerance/unacceptable toxicity. Each maintenance cycle is 28 days.
  Randomisation 2 is double-blind - participants and their treating clinicians will be blinded to maintenance allocation.
  Other Names: Revlimid; Ninlaro
  Arms: R2: Lenalidomide + ixazomib maintenance

SUMMARY:
Trial Title:

FiTNEss (UK-MRA Myeloma XIV) - Frailty-adjusted therapy in Transplant Non-Eligible patients with newly diagnosed Multiple Myeloma

Overview:

A phase III, multi-centre, randomised controlled trial to compare standard (reactive) and frailty-adjusted (adaptive) induction therapy delivery with the novel triplet ixazomib, lenalidomide and dexamethasone (IRD), and to compare maintenance lenalidomide (R) to lenalidomide plus ixazomib (R+I) in patients with newly diagnosed multiple myeloma not suitable for a stem cell transplant.

All participants receive induction treatment with ixazomib, lenalidomide and dexamethasone and are randomised on a 1:1 basis at trial entry to the use of frailty score-adjusted up-front dose reductions vs. standard up-front dosing followed by toxicity dependent reactive dose-modifications during therapy. Following 12 cycles of induction treatment participants alive and progression-free undergo a second randomisation on a 1:1 basis to maintenance treatment with lenalidomide plus placebo versus lenalidomide plus ixazomib. Participants and their treating physicians will be blinded to maintenance allocation.

Participant population:

* Newly diagnosed as having Multiple Myeloma (MM) according to the updated IMWG diagnostic criteria 2014 (see Appendix 1 for criteria)
* Not eligible for stem cell transplant
* Aged at least 18 years
* Able to provide written informed consent

Number of participants:

740 participants will be entered into the trial at Randomisation 1 (R1), with 478 participants at Randomisation 2 (R2).

Objectives:

The primary objectives of this study are to determine:

* Early treatment cessation (within 60 days of randomisation) for standard versus frailty-adjusted up-front dosing
* Progression-free survival (PFS, from maintenance randomisation) for lenalidomide + placebo (R) versus lenalidomide + ixazomib (R+I)

The secondary objectives of this study are to assess progression-free survival (PFS) for standard versus frailty-adjusted up-front dosing reductions, time to progression, time to 2nd PFS event (PFS2), overall survival (OS), survival after progression, deaths within 12 months of R1, overall response rate (ORR), attainment of ≥VGPR, attainment of MRD negativity, duration of response, time to improved response, time to next treatment, treatment compliance and total amount of therapy delivered, toxicity & safety including the incidence of SPMs, Quality of Life (QoL), cost effectiveness of standard versus frailty-adjusted up-front dosing of IRD and cost-effectiveness of R + I versus R.

Exploratory objectives are prospective validation of a novel frailty risk score (UK-MRA Myeloma Risk Profile - MRP), usefulness of Karnofsky Performance Status (PS), and association of molecular subgroups with response, PFS and OS.

ELIGIBILITY:
Eligibility criteria for Randomisation 1 (R1) Participants must meet all of the following inclusion criteria and none of the exclusion criteria.

Inclusion criteria for R1

1. Newly diagnosed as having MM according to the updated IMWG diagnostic criteria 2014 requiring treatment.
2. Not eligible for stem cell transplant.
3. Aged at least 18 years.
4. Meet all of the following blood criteria within 14 days before R1:

   Haematological:
   1. Absolute neutrophil count (ANC) ≥ 1 x 10^9/L. Unless the participant has a known/suspected diagnosis of familial or racial neutropenia in which case an ANC ≥ 0.75 x 10^9/L is allowed. The use of growth factor support is permitted.
   2. Platelet count ≥ 50 x 10^9/L, or, in the case of heavy bone marrow infiltration (≥ 50%) which in the opinion of the investigator is the cause of the thrombocytopenia and provided appropriate supportive measures and patient monitoring are in place, platelet count ≥ 30 x 10^9/L is permitted. Please note: Platelet transfusions are not allowed ≤ 3 days prior to randomisation in order to meet these values.
   3. Haemoglobin ≥ 80 g/L. The use of red blood cell transfusions is permitted.

      Biochemical:
   4. Total bilirubin ≤ 3 x upper limit of normal (ULN).
   5. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3 x ULN.
5. Meet the pregnancy prevention requirements:

   Female participants who:
   1. Are not of childbearing potential, OR
   2. If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form until 90 days after the last dose of study drug, OR
   3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilised (i.e. status post-vasectomy), must agree to one of the following:
   1. Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
   2. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

   Contraception for female and male participants must be in accordance with (and participants must consent to) the Celgene-approved Pregnancy Prevention Programme.

   If female and of childbearing potential, they must have a negative pregnancy test performed by a healthcare professional in accordance with the Celgene Pregnancy Prevention Programme.
6. Able to provide written informed consent.

Exclusion criteria for R1

1. Smouldering MM, MGUS, solitary plasmacytoma of bone, or extramedullary plasmacytoma (without evidence of MM).
2. Received previous treatment for MM, with the exception of local radiotherapy to relieve bone pain or spinal cord compression, prior bisphosphonate treatment, or corticosteroids as long as the total dose does not exceed the equivalent of 160 mg dexamethasone.
3. Known resistance, intolerance or sensitivity to any component of the planned therapies.
4. Prior or concurrent invasive malignancies except the following:

   * Adequately treated basal cell or squamous cell skin cancer;
   * Incidental finding of low grade (Gleason 3+3 or less) prostate cancer requiring no intervention;
   * Adequately treated carcinoma in situ of the breast or cervix no longer requiring medical or surgical intervention;
   * Any cancer from which the subject has been disease-free for at least 3 years.
5. Pregnant, lactating or breastfeeding female participants.
6. Major surgery within 14 days before randomisation. This would include surgical intervention for relief of cord compression but does not include vertebroplasty or kyphoplasty.
7. Systemic treatment, within 14 days before the first dose of ixazomib with strong CYP3A inducers (e.g. rifampicin, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
8. Any concomitant drug therapy which, in the opinion of the investigator, may lead to an unacceptable interaction with any of the agents ixazomib, lenalidomide, dexamethasone, and that cannot be safely stopped prior to trial entry. Full details of interactions can be found in the SPCs.
9. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of trial treatment, including difficulty swallowing.
10. ≥ Grade 2 peripheral neuropathy.
11. Known HIV positive or known hepatitis B surface antigen positive or hepatitis C antibody positive.
12. Active systemic infection.
13. Any other medical or psychiatric condition which, in the opinion of the investigator, contraindicates the participant's participation in this study.

Eligibility criteria for Randomisation 2 (R2) Participants must meet all of the following inclusion criteria and none of the exclusion criteria.

Inclusion criteria for R2

1. Randomised into the FiTNEss (Myeloma XIV) trial and received induction chemotherapy with ixazomib and lenalidomide continued for 12 cycles.
2. Achieved at least MR at the end of IRD induction according to the IMWG Uniform Response Criteria for Multiple Myeloma, with no evidence of progression prior to R2.
3. Meet all of the following blood criteria within 14 days before R2:

Haematological:

1. Absolute neutrophil count (ANC) ≥ 1 x 10^9/L. Unless the participant has a known/suspected diagnosis of familial or racial neutropenia in which case an ANC ≥ 0.75 x 10^9/L is allowed. The use of growth factor support is permitted.
2. Platelet count ≥ 50 x 10^9/L. Please note: Platelet transfusions are not allowed ≤ 3 days prior to randomisation in order to meet these values.
3. Haemoglobin ≥ 80 g/L. The use of red blood cell transfusions is permitted.

   Biochemical:
4. Total bilirubin ≤ 3 x upper limit of normal (ULN).
5. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3 x ULN.

Exclusion criteria for R2

1. Received any anti-myeloma therapy other than their randomised trial treatment, with the exception of local radiotherapy to relieve bone pain (in the absence of disease progression), or bisphosphonate treatment.
2. SD or disease progression according to the IMWG Uniform Response Criteria for Multiple Myeloma.
3. Known resistance, intolerance or sensitivity to ixazomib or lenalidomide that required cessation of either agent during induction.
4. Developed any malignancy since R1 except the following:

   * Adequately treated basal cell or squamous cell skin cancer;
   * Incidental finding of low grade (Gleason 3+3 or less) prostate cancer requiring no intervention;
   * Adequately treated carcinoma in situ of the breast or cervix no longer requiring medical or surgical intervention.
5. Pregnant, lactating or breastfeeding female participants.
6. Major surgery within 14 days before randomisation. This does not include vertebroplasty or kyphoplasty.
7. Systemic treatment, within 14 days before the first dose of ixazomib with strong CYP3A inducers (e.g. rifampicin, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
8. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of trial treatment, including difficulty swallowing.
9. ≥ Grade 2 peripheral neuropathy, or grade 1 with pain.
10. Known HIV positive or known hepatitis B surface antigen positive or hepatitis C antibody positive.
11. Active systemic infection.
12. Any other medical or psychiatric condition which, in the opinion of the investigator, contraindicates the participant's continued participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Randomisation 1: Number of participants with early treatment cessation | Within 60 days of Randomisation 1
  Early treatment cessation is defined as a binary endpoint. Participants will be defined to have experienced an event if they die, progress, or are withdrawn from treatment (by a treating clinician) or withdraw consent for trial treatment, within 60 days of Randomisation 1.
Randomisation 2: Progression-free survival (PFS-R2) | The time from the date of Randomisation 2 to the date of first documented evidence of disease progression or death from any cause, up to 120 months
  PFS-R2 is defined as the time from Randomisation 2 to the time of first documented evidence of disease progression or death from any cause. Individuals who are lost to follow-up or progression-free at the time of analysis will be censored at their last known date to be alive and progression-free. Disease progression is defined according to the IMWG Uniform Response Criteria for Multiple Myeloma.

SECONDARY OUTCOMES:
Progression-free survival (PFS-R1) | The time from the date of Randomisation 1 to the date of first documented evidence of disease progression or death from any cause, up to 120 months
  PFS-R1 is defined as the time from R1 to the time of first documented evidence of disease progression or death from any cause. Individuals who are lost to follow-up or progression-free at the time of analysis will be censored at their last known date to be alive and progression-free. Disease progression is defined according to the IMWG Uniform Response Criteria for Multiple Myeloma.
Time to disease progression | The time from the date of randomisation to the date of first documented evidence of disease progression, up to 120 months
  Time to disease progression is defined for both Randomisation 1 and Randomisation 2 as the time from randomisation to the date of first documented evidence of disease progression. Participants who die prior to documentation of disease progression will be censored in the analysis at their date of death. Participants not reaching disease progression at the time of analysis will be censored at the last date known to be progression-free. Participants dying from causes not primarily due to progression will also be censored.
Progression-free survival two (PFS2) | The time from the date of randomisation to the date of the second documented disease progression, up to 120 months
  For both Randomisation 1 and Randomisation 2, progression-free survival two is defined as the time from randomisation to the time of the second documented disease progression. Individuals who are lost to follow-up or second progression-free at the time of analysis will be censored at their last known date to be alive and second progression-free.
Overall survival (OS) | The time from the date of randomisation to the date of death from any cause, up to 120 months
  Overall survival is defined separately for each randomisation. In each case it is the time from randomisation to the time of death from any cause. Individuals who are lost to follow-up or still alive at the time of analysis will be censored at their last known date to be alive.
Survival after progression | The date of first documented evidence of disease progression to the date of death from any cause, up to 120 months
  Survival after progression is defined from the date of first documented evidence of disease progression to the date of death from any cause. Individuals who are lost to follow-up or alive at the time of analysis will be censored at their last known date to be alive following their first documented evidence of disease progression.
Deaths within 12 months of Randomisation 1 (R1) | Within 12 months of Randomisation 1
  Deaths within 12 months of Randomisation 1 is defined as a binary endpoint. Participants will be defined to have experienced an event if they die within 12 months of Randomisation 1.
Overall response rate (ORR) | From the date of Randomisation 1 to the end of 12 cycles of induction treatment (each induction cycle is 28 days)
  Overall response rate is defined as a categorical outcome consisting of whether a participant had Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD) or Progressive Disease (PD) at the end of induction according to the IMWG Uniform Response Criteria for Multiple Myeloma.
Attainment of ≥VGPR | From the date of Randomisation 1 to the end of 12 cycles of induction treatment (each induction cycle is 28 days)
  Attainment of ≥VGPR is defined as a binary outcome of whether a participant had ≥VGPR (VGPR, CR, sCR) or <VGPR (PR, MR, SD, PD) at the end of induction, according to the IMWG Uniform Response Criteria for Multiple Myeloma.
Attainment of Minimal Residual Disease (MRD) negativity | From the date of Randomisation 1 to the end of 12 cycles of induction treatment (each induction cycle is 28 days); and 12 months after the date of Randomisation 2
  Attainment of Minimal Residual Disease (MRD) negativity is defined as a binary endpoint. MRD negativity will be determined at the end of induction therapy and 12 months post Randomisation 2 according to the IMWG MRD criteria.
Duration of response (DoR) | The time from the date of the first observation of response ≥ Partial Response following Randomisation 1, to the date of first documented evidence of disease progression or death confirmed related to progression, up to 120 months
  Duration of response is defined as the time from the first observation of response ≥ Partial Response (PR), following Randomisation 1, to the time of first documented evidence of disease progression or death confirmed related to progression. Individuals who are lost to follow-up, or still alive and progression-free at the time of analysis will be censored at their last known date to be alive and progression-free. Individuals whose cause of death is unrelated to disease progression will be censored at their date of death.
Time to improved response | The time from the date of Randomisation 2 to the date the response category is first improved, up to 120 months
  Time to improved response is defined as the time from the date of Randomisation 2 to the date the response category is first improved based on the Modified International Uniform Response Criteria for Multiple Myeloma. Subjects without any improvement of the baseline status at Randomisation 2 will be censored at the last date of response assessment.
Time to next treatment | The time from the date of Randomisation 1 to the start date of the next line of treatment or death from any cause, up to 120 months
  Time to next treatment is defined as the time from Randomisation 1 to the start date of the next line of treatment or death from any cause.
Treatment compliance and total amount of therapy delivered | Number of induction and maintenance cycles a participant received (each cycle of induction or maintenance is 28 days), until disease progression, up to 120 months
  In the first instance treatment compliance is defined as a binary outcome i.e. did the participant receive 12 cycles of induction treatment. The total amount of therapy delivered will be first defined as the number of induction and maintenance cycles which the participant received. This may be extended to consider the percentage of protocol dose delivered. For each treatment (ixazomib, lenalidomide, dexamethasone) this will be defined as the total dose received in a cycle compared to the total dose the participant should have received in the cycle without modifications, averaged across all cycles of treatment.
Incidence of treatment-emergent adverse events (Toxicity and safety, including incidence of second malignancies) | Baseline, end of each induction cycle (each induction cycle is 28 days), end of each maintenance cycle (each maintenance cycle is 28 days), until disease progression, up to 120 months
  Toxicity & safety, including incidence of second malignancies Toxicity and safety will be reported based on the adverse events, as graded by CTCAE V5 and determined by routine clinical assessments at each centre. The number of SAEs will be reported according to MedDRA System Organ Class. All second primary malignancies will be reported based on information collected on the Case Report Form.
EORTC QLQ-C30_questionnaire | Randomisation 1; after cycles 2, 4, 6 and 12 of induction treatment (each induction cycle is 28 days); after cycles 6 and 12 of maintenance treatment (each maintenance cycle is 28 days)
  European Organization for the Research & Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) is used to measure patient-assessed quality of life (QoL) at R1, after cycles 2, 4, 6 & 12 of induction, and after cycles 6 and 12 of maintenance (all cycles are 28 days).
  The QLQ-C30 comprises multi-item scales & single-item measures: 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, pain, nausea & vomiting), a global health status/QoL scale, & 6 single items assessing additional symptoms (dyspnoea, loss of appetite, insomnia, constipation & diarrhoea). All scales & single-item measures range in score from 0 to 100. A high scale score represents a higher response level: a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high quality of life, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
EORTC QLQ-MY20_questionnaire | Randomisation 1; after cycles 2, 4, 6 and 12 of induction treatment (each induction cycle is 28 days); after cycles 6 and 12 of maintenance treatment (each maintenance cycle is 28 days)
  The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Multiple Myeloma Module (EORTC QLQ-MY20) is used to measure patient-assessed quality of life (QoL) at Randomisation 1, after cycles 2, 4, 6 and 12 of induction treatment (each induction cycle is 28 days), and after cycles 6 and 12 of maintenance treatment (each maintenance cycle is 28 days).
  The EORTC QLQ-MY20 comprises 20 questions that address four myeloma-specific QoL domains: Disease Symptoms, Side Effects of Treatment, Future Perspectives, and Body Image. Disease Symptoms, Side Effects of Treatment, and Future Perspectives are all multi-item scales, and Body Image is a single-item scale. Domain scores are averaged and transformed linearly to a score ranging from 0-100. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.
EQ-5D-3L_questionnaire | Randomisation 1; after cycles 2, 4, 6 and 12 of induction treatment (each induction cycle is 28 days); after cycles 6 and 12 of maintenance treatment (each maintenance cycle is 28 days)
  The EuroQol 5 Dimension 3 Level questionnaire (EQ-5D-3L) will be used to measure participant-assessed quality of life at Randomisation 1, after cycles 2, 4, 6 and 12 of induction treatment (each induction cycle is 28 days), and after cycles 6 and 12 of maintenance treatment (each maintenance cycle is 28 days).
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

OTHER OUTCOMES:
Novel frailty risk score (UK-MRA MRP)_composite measure | Through study completion, up to 120 months
  The prospective validation of a novel frailty risk score (UK Myeloma Research Alliance Myeloma Risk Profile (UK-MRA MRP)) will use the following measurements at baseline to categorise individuals into fit, intermediate-fitness and frail using the UK-MRA MRP:
  * C-Reactive Protein (CRP),
  * Age,
  * Performance status on Eastern Cooperative Oncology Group (ECOG) scale (scoring from 0 to 5, with 0 - fully active and 5 = dead) and
  * Score on Revised International Staging System for Multiple Myeloma scale (ISS). The ISS score categorises newly-diagnosed myeloma patients into three groups (I, II, or III) depending on expected prognosis/overall survival based on measurements of serum beta-2 microglobulin and serum albumin.
Usefulness of Karnofsky PS_composite measure | Through study completion, up to 120 months
  The Karnofsky Performance Status will be contrasted with the Eastern Cooperative Oncology Group (ECOG) Performance Status to consider whether it can appropriately measure the performance status of patients with multiple myeloma.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Cook, MD, Principal Investigator — University of Leeds; Graham Jackson, MD, Principal Investigator — Freeman Hospital, Newcastle-Upon-Tyne
Locations (110):
- United Kingdom (110):
  - Aberdeen Royal Infirmary, Aberdeen
  - Nevill Hall Hospital, Abergavenny
  - Wrightington Hosptial, Appley Bridge
  - Ysbyty Gwynedd, Bangor
  - North Devon District Hospital, Barnstaple
  - Furness General Hospital, Barrow in Furness
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bolton Hospital, Bolton
  - Pilgrim Hospital, Boston
  - Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Bristol Haematology and Oncology Centre, Bristol
  - Southmead Hospital, Bristol
  - Queen's Hospital, Burton-on-Trent
  - Kent and Canterbury Hospital, Canterbury
  - Chelmsford & Essex Hospital, Chelmsford
  - Cheltenham General Hospital, Cheltenham
  - Countess of Chester Hospital, Chester
  - St Richard's Hospital, Chichester
  - Colchester General Hospital, Colchester
  - University Hospital Coventry, Coventry
  - Croydon University Hospital, Croydon
  - Royal Derby Hospital, Derby
  - Dorset County Hospital, Dorchester
  - Russells Hall Hospital, Dudley
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Medway Maritime Hospital, Gillingham
  - Gloucestershire Royal Hospital, Gloucester
  - Grantham and District Hospital, Grantham
  - Diana Princess of Wales Hospital, Grimsby
  - Royal Surrey County Hospital, Guildford
  - Calderdale Royal Hospital, Halifax
  - Harrogate District Hospital, Harrogate
  - Withybush General Hospital, Haverfordwest
  - Hereford County Hospital, Hereford
  - Huddersfield Royal Infirmary, Huddersfield
  - Castle Hill Hospital, Hull
  - Raigmore Hospital, Inverness
  - Ipswich Hospital, Ipswich
  - Airedale Hospital, Keighley
  - Westmorland General Hospital, Kendal
  - Kettering General Hospital, Kettering
  - Kidderminster Hospital & Treatment Centre, Kidderminster
  - Victoria Hospital, Kirkcaldy
  - Royal Lancaster Infirmary, Lancaster
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Aintree University Hospital, Liverpool
  - Royal Liverpool Hospital, Liverpool
  - Guy's Hospital, London
  - King's College Hospital, London
  - Queen Elizabeth Hospital Greenwich, London
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - University Hospital Lewisham, London
  - Maidstone Hospital, Maidstone
  - Manchester Royal Infirmary, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - Royal Gwent Hospital, Newport
  - North Tyneside General Hospital, North Shields
  - Nottingham City Hospital, Nottingham
  - Royal Oldham Hospital, Oldham
  - Princess Royal University Hospital, Orpington
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Whiston Hospital, Prescot
  - Royal Preston Hospital, Preston
  - Royal Berkshire Hospital, Reading
  - Alexandra Hospital, Redditch
  - Glan Clwyd Hospital, Rhyl
  - Queen's Hospital, Romford
  - Tunbridge Wells Hospital, Royal Tunbridge Wells
  - Salford Royal Hospital, Salford
  - Salisbury District Hospital, Salisbury
  - Scarborough General Hospital, Scarborough
  - Scunthorpe General Hospital, Scunthorpe
  - Royal Hallamshire Hospital, Sheffield
  - Royal Shrewsbury Hospital, Shrewsbury
  - Southampton General Hospital, Southampton
  - St Helens Hospital, St Helens
  - Stafford County Hospital, Stafford
  - Stepping Hill Hospital, Stockport
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - Good Hope Hospital, Sutton Coldfield
  - Singleton Hospital, Swansea
  - St George's Hospital, Tooting
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Hillingdon Hospital, Uxbridge
  - Pinderfields General Hospital, Wakefield
  - Warwick Hospital, Warwick
  - Sandwell General Hospital, West Bromwich
  - Royal Albert Edward Infirmary, Wigan
  - Royal Hampshire County Hospital, Winchester
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - Worthing Hospital, Worthing
  - Wrexham Maelor Hospital, Wrexham
  - York Hospital, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coulson AB, Royle KL, Pawlyn C, Cairns DA, Hockaday A, Bird J, Bowcock S, Kaiser M, de Tute R, Rabin N, Boyd K, Jones J, Parrish C, Gardner H, Meads D, Dawkins B, Olivier C, Henderson R, Best P, Owen R, Jenner M, Kishore B, Drayson M, Jackson G, Cook G. Frailty-adjusted therapy in Transplant Non-Eligible patients with newly diagnosed Multiple Myeloma (FiTNEss (UK-MRA Myeloma XIV Trial)): a study protocol for a randomised phase III trial. BMJ Open. 2022 Jun 2;12(6):e056147. doi: 10.1136/bmjopen-2021-056147. PMID 35654466